CLINICAL TRIAL: NCT00004781
Title: Oral Manifestations of Human Immunodeficiency Virus Infection in High Risk Groups
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Collaborators: Columbia University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11861; CU-SDOS-5059
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-02

CONDITIONS: HIV Infections; Candidiasis, Oral
Keywords: HIV-associated candidiasis; candidiasis; disease-related problem/condition; fungal infection; immunologic disorders and infectious disorders; infection; rare disease
MeSH Terms: conditions — HIV Infections; Candidiasis, Oral; Candidiasis; Mycoses; Immune System Diseases; Communicable Diseases; Infections; Rare Diseases

SUMMARY:
OBJECTIVES: I. Evaluate the development of oral manifestations of human immunodeficiency virus infection in relationship to the onset of immunologic alterations and systemic symptoms in different risk groups: gay/bisexual men, male intravenous drug users, and female intravenous drug users.

II. Evaluate the immune and inflammatory response to periodontal and other microbial pathogens.

III. Evaluate the bacterial species infecting the oral cavity in patients in these risk groups.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients undergo a periodontal assessment every 6 months until medically unable to continue. The oral/dental exam includes saliva and gingival crevicular fluid analysis and, as indicated, oral photographs.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Human immunodeficiency virus infection (HIV) seropositive or seronegative At risk for HIV, i.e.: Gay/bisexual men Male intravenous drug users Female intravenous drug users No acquired immunodeficiency syndrome Currently enrolled in Columbia Presbyterian Medical Center protocol "The Natural History and Progression of HIV Infection"

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 1989-09

CONTACTS AND LOCATIONS:
Overall Officials: Ira B. Lamster, Study Chair — Columbia University